CLINICAL TRIAL: NCT04016298
Title: Validation of Bladder Health Instrument for Evaluation in Women
Acronym: VIEW
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Collaborators: University of California, San Diego (Other); University of Pennsylvania (Other); Yale University (Other); University of Michigan (Other); University of Illinois at Chicago (Other); Loyola University Chicago (Other); University of Alabama at Birmingham (Other); Washington University School of Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00032238
Record Dates: First submitted 2019-07-05; First posted 2019-07-11 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Lower Urinary Tract Symptoms
Keywords: Bladder Health; LUTS; PLUS; VIEW
MeSH Terms: conditions — Lower Urinary Tract Symptoms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Prevention of Lower Urinary Symptoms (PLUS) Research Consortium is working to optimize prevention of lower urinary tract symptoms (LUTS) in women and adolescent females across their life spans. The ability to measure bladder health and key risk and protective factors is crucial to the PLUS mission. To describe and measure the spectrum of bladder health in diverse populations, researchers need a valid and reliable instrument. To date, the Consortium's work on design of a bladder health instrument has been a culmination of expert opinion, information from focus groups, and incorporation of previously validated items and language where appropriate, along with cognitive interviews of participants from the general public. The next step in the consortium's work is to prospectively collect data to test and validate bladder health instrument (BHI) items for inclusion in a final bladder health scale (BHS) that can assess the full range of bladder health of women. This will be through a combination of general population recruitment for completing mailed surveys, clinical population recruitment for completing surveys and an in-person evaluation, and postpartum women.

ELIGIBILITY:
Inclusion Criteria:

* Community dwelling
* Age ≥18 years old
* Female sex assigned at birth
* Fluent in written and spoken English
* Able to read and provide informed consent

Exclusion Criteria:

* Institutional living arrangement, e.g., skilled nursing, long term care or rehabilitation center
* Physical or mental condition that would prohibit self-administration of questionnaire either electronically or using paper and pencil (e.g., dementia/cognitive impairment/blindness/severe arthritis).

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The BHI is intended for use in the general US population and it is critical that the BHI validation include individuals who meet these criteria. The goal is to include women over the age of 18 that meet the inclusion criteria. It is our hope to get a broad spectrum of women with varying degrees of bladder health, age, race, and community.
Sampling Method: Probability Sample
Enrollment: 1222 (Actual)
Dates: Start 2019-07-31 (Actual); Primary Completion 2022-05-25 (Actual); Study Completion 2022-05-25 (Actual)

PRIMARY OUTCOMES:
Bladder Health Instrument | Will be assessed throughout the duration of study, an average of one year.
  Multi-item measurement is used to assess the range of bladder health dimensions as defined by the model of bladder health adopted by the PLUS consortium. It is anticipated that the self-administeredBHI instrument (PAPI or CASI) will consist of approximately 85 items: 53-67 are items all respondents will be asked to answer, and 48 are asked only of women who self-identify as experiencing a specific LUTS. The items cover the range of bladder health dimensions specified by our model.

CONTACTS AND LOCATIONS:
Overall Officials: Emily Lukacz, MD, Principal Investigator — University of California, San Diego
Locations (8):
- United States (8):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - University of California, San Diego, San Diego, California
  - Yale University, New Haven, Connecticut
  - Loyola University Chicago, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - University of Minnesota, Minneapolis, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Lukacz ES, Bavendam TG, Berry A, Fok CS, Gahagan S, Goode PS, Hardacker CT, Hebert-Beirne J, Lewis CE, Lewis J, Low LK, Lowder JL, Palmer MH, Smith AL, Brady SS. A Novel Research Definition of Bladder Health in Women and Girls: Implications for Research and Public Health Promotion. J Womens Health (Larchmt). 2018 Aug;27(8):974-981. doi: 10.1089/jwh.2017.6786. Epub 2018 May 24. PMID 29792542
- [Background] Brady SS, Bavendam TG, Berry A, Fok CS, Gahagan S, Goode PS, Hardacker CT, Hebert-Beirne J, Lewis CE, Lewis JB, Kane Low L, Lowder JL, Palmer MH, Wyman JF, Lukacz ES; Prevention of Lower Urinary Tract Symptoms (PLUS) Research Consortium. The Prevention of Lower Urinary Tract Symptoms (PLUS) in girls and women: Developing a conceptual framework for a prevention research agenda. Neurourol Urodyn. 2018 Nov;37(8):2951-2964. doi: 10.1002/nau.23787. Epub 2018 Aug 22. PMID 30136299
- [Background] Bandilla W, Bosnjak M, Altdorfer P. Survey Administration Effects?: A Comparison of Web-Based and Traditional Written Self-Administered Surveys Using the ISSP Environment Module. Soc Sci Comput Rev. 2003;21(2):235-243. doi:10.1177/0894439303021002009.
- [Background] Dillman DA, Sangster RL, Tarnai J, Rockwood TH. Understanding differences in people's answers to telephone and mail surveys. New Dir Eval. 1996;1996(70):45-61. doi:10.1002/ev.1034.
- [Background] Vernon SW, Tiro JA, Vojvodic RW, Coan S, Diamond PM, Greisinger A, Fernandez ME. Reliability and validity of a questionnaire to measure colorectal cancer screening behaviors: does mode of survey administration matter? Cancer Epidemiol Biomarkers Prev. 2008 Apr;17(4):758-67. doi: 10.1158/1055-9965.EPI-07-2855. Epub 2008 Apr 1. PMID 18381467
- [Background] Schwarz N, Strack F, Hippler H, Bishop G. The impact of administration mode on response effects in survey measurement. Jobe JB, Loftus EF, eds. Appl Cogn Psychol. 1991;5(3):193-212. doi:10.1002/acp.2350050304.
- [Background] Cronbach L. Coefficient alpha and the internal structure of tests. Psychometrika. 1951;16(3):297-334. doi:10.1007/BF02310555.
- [Background] Swartz RJ, de Moor C, Cook KF, Fouladi RT, Basen-Engquist K, Eng C, Carmack Taylor CL. Mode effects in the center for epidemiologic studies depression (CES-D) scale: personal digital assistant vs. paper and pencil administration. Qual Life Res. 2007 Jun;16(5):803-13. doi: 10.1007/s11136-006-9158-0. Epub 2007 Feb 13. PMID 17295102
- [Background] Messick S. The interplay of evidence and consequences in the validation of performance assessments. ETS Res Rep Ser. 1992;1992(1):i-42. doi:10.1002/j.2333-8504.1992.tb01470.x.
- [Background] Kane MT. Validating the Interpretations and Uses of Test Scores. J Educ Meas. 2013;50(1):1-73. doi:10.1111/jedm.12000.
- [Background] Hawkins M, Elsworth GR, Osborne RH. Application of validity theory and methodology to patient-reported outcome measures (PROMs): building an argument for validity. Qual Life Res. 2018 Jul;27(7):1695-1710. doi: 10.1007/s11136-018-1815-6. Epub 2018 Feb 20. PMID 29464456
- [Background] American Educational Research Association. Standards for Educational and Psychological Testing. (Association AP, Education NC on M in, (U.S.) JC on S for E and PT, eds.). Washington, DC: Washington, DC : American Educational Research Association; 2014.
- [Background] Streiner D. Health Measurement Scales : A Practical Guide to Their Development and Use. Fifth edit. (Norman GR, Cairney J, ebrary I, eds.). New York, New York: New York, New York : Oxford University Press; 2015.
- [Background] Messick S. VALIDITY. Educ Test Serv Res Rep Ser. 1987;1987(2):i-208. doi:10.1002/j.2330-8516.1987.tb00244.x.
- [Background] CAMPBELL DT, FISKE DW. Convergent and discriminant validation by the multitrait-multimethod matrix. Psychol Bull. 1959 Mar;56(2):81-105. No abstract available. PMID 13634291
- [Background] Martin JA, Hamilton BE, Osterman MJK, Driscoll AK, Drake P. Births: Final Data for 2017. Natl Vital Stat Rep. 2018 Nov;67(8):1-50. PMID 30707672
- [Background] Chin HB, Baird DD, McConnaughey DR, Weinberg CR, Wilcox AJ, Jukic AM. Long-term Recall of Pregnancy-related Events. Epidemiology. 2017 Jul;28(4):575-579. doi: 10.1097/EDE.0000000000000660. PMID 28346268
- [Background] McHorney CA, Ware JE Jr, Raczek AE. The MOS 36-Item Short-Form Health Survey (SF-36): II. Psychometric and clinical tests of validity in measuring physical and mental health constructs. Med Care. 1993 Mar;31(3):247-63. doi: 10.1097/00005650-199303000-00006. PMID 8450681
- [Background] Kelleher CJ, Cardozo LD, Khullar V, Salvatore S. A new questionnaire to assess the quality of life of urinary incontinent women. Br J Obstet Gynaecol. 1997 Dec;104(12):1374-9. doi: 10.1111/j.1471-0528.1997.tb11006.x. PMID 9422015
- [Background] Naughton MJ, Donovan J, Badia X, Corcos J, Gotoh M, Kelleher C, Lukacs B, Shaw C. Symptom severity and QOL scales for urinary incontinence. Gastroenterology. 2004 Jan;126(1 Suppl 1):S114-23. doi: 10.1053/j.gastro.2003.10.059. PMID 14978647
- [Background] Barber MD, Walters MD, Bump RC. Short forms of two condition-specific quality-of-life questionnaires for women with pelvic floor disorders (PFDI-20 and PFIQ-7). Am J Obstet Gynecol. 2005 Jul;193(1):103-13. doi: 10.1016/j.ajog.2004.12.025. PMID 16021067
- [Background] Jackson S, Donovan J, Brookes S, Eckford S, Swithinbank L, Abrams P. The Bristol Female Lower Urinary Tract Symptoms questionnaire: development and psychometric testing. Br J Urol. 1996 Jun;77(6):805-12. doi: 10.1046/j.1464-410x.1996.00186.x. PMID 8705212
- [Background] Miller JM, Ashton-Miller JA, Delancey JO. Quantification of cough-related urine loss using the paper towel test. Obstet Gynecol. 1998 May;91(5 Pt 1):705-9. doi: 10.1016/s0029-7844(98)00045-3. PMID 9572215
- [Background] Gorsuch RL. Common Factor Analysis versus Component Analysis: Some Well and Little Known Facts. Multivariate Behav Res. 1990 Jan 1;25(1):33-9. doi: 10.1207/s15327906mbr2501_3. No abstract available. PMID 26741966
- [Derived] Rickey LM, Mueller ER, Newman DK, Markland AD, Falke C, Rudser K, Smith AL, Mueller MG, Lowder JL, Lukacz ES; Prevention of Lower Urinary Tract Symptoms (PLUS) Research Consortium. Reliability of Uroflowmetry Pattern Interpretation in Adult Women. Neurourol Urodyn. 2024 Nov;43(8):2084-2092. doi: 10.1002/nau.25584. Epub 2024 Sep 12. PMID 39264028
- [Derived] Constantine ML, Rockwood TH, Rickey LM, Bavendam T, Low LK, Lowder JL, Markland AD, McGwin G, Mueller ER, Newman DK, Putnam S, Rudser K, Smith AL, Stapleton AE, Miller JM, Lukacz ES; of the Prevention of Lower Urinary Tract Symptoms (PLUS) Research Consortium. Validation of bladder health scales and function indices for women's research. Am J Obstet Gynecol. 2023 May;228(5):566.e1-566.e14. doi: 10.1016/j.ajog.2022.12.319. Epub 2022 Dec 31. PMID 36596439
- [Derived] Lukacz ES, Constantine ML, Kane Low L, Lowder JL, Markland AD, Mueller ER, Newman DK, Rickey LM, Rockwood T, Rudser K; Prevention of Lower Urinary Tract Symptoms (PLUS) Research Consortium. Rationale and design of the validation of bladder health instrument for evaluation in women (VIEW) protocol. BMC Womens Health. 2021 Jan 7;21(1):18. doi: 10.1186/s12905-020-01136-w. PMID 33413284